CLINICAL TRIAL: NCT05234437
Title: A Phase IIb, Multicentre, Open Label Study to Evaluate the Effectiveness, Safety and Tolerability of Intratumoural Tigilanol Tiglate in Adult Participants With Stage IIIB to IV M1c Melanoma
Brief Title: A Trial of Intratumoural Tigilanol Tiglate in Adult Participants With Stage IIIB to IV M1c Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Patient Recruitment Rates
Sponsor: QBiotics Group Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QB46C-H04; U1111-1258-4085 (Registry Identifier: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2022-01-11; First posted 2022-02-10 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-10

CONDITIONS: Melanoma
Keywords: Melanoma; Intratumoural; Epoxytigilane; Tigilanol Tiglate
MeSH Terms: conditions — Melanoma | interventions — EBC-46

STUDY DESIGN:
Intervention Model Description: Open-label multicentre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm open label (Experimental): Single or multiple Intratumoural treatment of tigilanol tiglate at 3.6mg/m2 given at a minimum of 28-day intervals.
  Interventions: Drug: tigilanol tiglate

INTERVENTIONS:
Drug: tigilanol tiglate — Single or multiple Intratumoural treatments of tigilanol tiglate up to a fixed dose level of 3.6mg/m2.
  Tigilanol tiglate is a novel, short-chain diterpene ester in early clinical development for local treatment of a wide range of solid tumours.
  Other Names: EBC-46

SUMMARY:
A phase IIb, multicentre, open label study to evaluate the effectiveness, safety, and tolerability of intratumoural tigilanol tiglate in adult participants with Stage IIIB to IV M1c melanoma

DETAILED DESCRIPTION:
Primary Objective

1. To evaluate the tumour responses of both injected and non injected tumours following treatment with intratumoural injections of tigilanol tiglate into one or more tumours (according to RECIST v1.1); and
2. To assess the tumour ablation rate following treatments with intratumoural injections of tigilanol tiglate.

Secondary Objectives

1. To assess the tumour recurrence rate at injected tumour site(s);
2. To assess the safety and tolerability of intratumoural injections of tigilanol tiglate;
3. To assess the degree of wound healing at injection sites; and
4. To evaluate disease control by looking at Progression Free Survival (PFS) in melanoma participants receiving tigilanol tiglate injections over 36 months.

Exploratory Objectives

1. To evaluate Overall Survival (OS) in melanoma participants receiving tigilanol tiglate injections over 36 months;
2. To assess the tumour microenvironment by looking at the degree of immune cell infiltration in non-injected tumours; and
3. To assess the Quality of Life (QoL) in melanoma participants receiving tigilanol tiglate injections.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for study participation if they meet ALL the following criteria:

  1. Are willing and able to provide written informed consent for the study prior to any protocol-required procedures and to comply with all study requirements. (Note: If a participant is unable to provide written informed consent, a legally acceptable representative may provide consent on their behalf).
  2. Are ≥ 18 years of age.
  3. Have a histologically confirmed diagnosis of melanoma that is Stage IIIB to IV M1c (AJCC 8th Ed.). These will be participants who are naïve to systemic therapy (i.e., not suitable for or have refused immunotherapy or targeted therapy), as well as participants who have progressed on a prior line of systemic therapy.
  4. Have measurable disease per RECIST v1.1 including cutaneous, subcutaneous, or nodal tumours consisting of ≥ 1 target tumours accessible and amenable to intratumoural injection that can be accurately measured by contrast enhanced CT as assessed by the Investigator's local site radiology.
  5. Are willing to undergo biopsy sampling of tumour(s).
  6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
  7. Have life expectancy of more than 12 weeks.
  8. Female participants of childbearing potential must have a negative serum β-HCG pregnancy test at Screening (within 14 days prior to commencement of study drug administration), must be willing to use adequate highly effective contraception 28 days prior to commencement of study drug administration and throughout the study up to 30 days after the last study drug administration, and must not be breastfeeding.
  9. Male participants with a potentially fertile partner are eligible if they have had a vasectomy or are willing to use adequate contraception and agree not donate sperm from commencement of study drug administration and throughout the study up to 30 days after the last study drug administration.

Exclusion Criteria:

* Participants will be excluded from study participation if they meet ANY of the following criteria:

  1. Are planning to receive intratumoural treatment or radiotherapy to any of the intended tumours for injection, or systemic therapy within 4 weeks prior to Screening, or during treatment with tigilanol tiglate.
  2. Have a tumour intended for treatment that is immediately adjacent to, or with infiltration into, any major artery or vein (e.g., if the tumour for injection is located adjacent to the jugular vein).
  3. Have a tumour intended for treatment located in an area where post-injection swelling could compromise the airway.
  4. Have had any previous intervention in the area of the intended tumour in proximity of the airway (e.g., radiation therapy to the area such that tracking of the injected fluid may be unpredictable and could lead to airway swelling).
  5. Have a histologically confirmed diagnosis of uveal melanoma as the only intended target tumour.
  6. Female participants that have a positive urine pregnancy test within 72 hours prior to the administration of study treatment(s) are not permitted to receive treatment (Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required).
  7. Participants who have received other investigational agents, have participated in a study of an investigational agent or have used an investigational device must undergo a 4-week wash-out period prior to Screening. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks after the last dose of the previous investigational agent. They must have recovered from all AEs due to previous therapies to ≤ Grade 1 at baseline visit, except participants who have experienced endocrine immune-related AEs. (Note: If a participant received major surgery, they must have recovered adequately from the morbidity and/or complications from the intervention prior to starting study treatment).
  8. Have known, current or history of central nervous system metastases, active cerebral metastasis and/or carcinomatous meningitis.
  9. Have any bleeding diathesis or coagulopathy that would make intratumoural injection or biopsy unsafe.
  10. Have significant peripheral vascular disease (e.g., participants who have claudication at rest) with accessible tumours intended for injection that are located in their extremities.
  11. Have a history of allergic reactions or severe hypersensitivity (Grade ≥ 3) attributed to tigilanol tiglate or compounds of similar chemical or biologic composition to tigilanol tiglate or any of its excipients or other agents used in the study.
  12. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
  13. In the opinion of the treating Investigator, the participant is an inappropriate candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Tumour Responses | 36 months
  - To evaluate the tumour responses of both injected and non injected tumours following treatment with intratumoural injections of tigilanol tiglate into one or more tumours (long term tumour response according to RECIST v1.1 criteria).
Tumour Ablation | 36 months
  - To assess the tumour ablation rate following treatment(s) with intratumoural injections of tigilanol tiglate.

SECONDARY OUTCOMES:
Tumour Recurrence Rate | 36 months
  - To assess the tumour recurrence rate at injected tumour site(s)
Safety and Tolerability | 36 months
  Total number of Adverse Events and Serious Adverse Events. Number of Adverse Events and Serious Adverse Events deemed related to tigilanol tiglate.
Wound Healing | 28 days
  - To assess the degree of wound healing at injection site(s) using a specifically designed Injection Site Assessment Worksheet, observed at 14 and 28 days post treatment.
Progression Free Survival (PFS) | 36 months
  - To evaluate disease control by looking at Progression Free Survival (PFS) in melanoma participants receiving tigilanol tiglate injections over 36 months

OTHER OUTCOMES:
Overall Survival (OS) | 36 months
  - To evaluate Overall Survival (OS) in melanoma participants receiving tigilanol tiglate injections
Tumour Microenvironment | 28 days
  - To assess the tumour microenvironment by looking at the degree of immune cell infiltration in non-injected tumours
Quality of Life (QoL) | 36 months
  QoL assessment using the Functional Assessment of Cancer Therapy - Melanoma (FACT-M) questionnaire at screening and at 6-monthly intervals until the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof. Robyn Saw, MBBS FRACS MS, Principal Investigator — Melanoma Institute Australia; Dr Megan Lyle, BMed FRACP, Principal Investigator — Cairns and Hinterland Hospital and Health Service; A/Professor Victoria Atkinson, Principal Investigator — Metro South Hospital and Health Service via Princess Alexandra Hospital
Locations (3):
- Australia (3):
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Cairns and Hinterland Hospital and Health Service, Cairns, Queensland
  - Metro South Hospital and Health Service via Princess Alexandra Hospital, Woolloongabba, Queensland